CLINICAL TRIAL: NCT01395823
Title: Safety and Effects of Supplementation With Ergocalciferol on Erythropoietin Dosing in Hemodialysis Patients: A Randomized Clinical Trial
Brief Title: Safety and Effects of Supplementation With Ergocalciferol on Erythropoietin Dosing in Hemodialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dialysis Clinic, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DCI-0002
Record Dates: First submitted 2011-07-14; First posted 2011-07-18 (Estimated); Results first posted 2016-03-14 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-02

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Vitamin D; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ergocalciferol supplementation (Other)
  Interventions: Dietary Supplement: ergocalciferol supplementation
- placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: ergocalciferol supplementation — 50,000 IU given either weekly; weekly for 3 months then monthly for 3 months; monthly
  Other Names: vitamin D, D2
  Arms: ergocalciferol supplementation
Other: placebo — placebo pill given weekly, weekly for 3 months then monthly for 3 months; monthly
  Other Names: sugar pill
  Arms: placebo

SUMMARY:
A few studies have reported erythropoiesis-stimulating agent (ESA) doses before and after 25D supplementation, but only one of these is a prospective clinical trial, and it is a small, single center study lacking a control arm. The investigators propose to conduct a double blind, randomized, placebo controlled clinical trial of ergocalciferol supplementation to confirm safety and determine effects on Erythropoietin (EPO) dosing, active D dosing, and mineral metabolic parameters in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients treated with thrice weekly in-center hemodialysis (HD) for more than 90 days.
2. Treated with EPO for at least 90 days. The mode of administration, intravenous (IV) or subcutaneous (SC), must remain the same for 90 days prior to enrollment.
3. The method by which EPO is prescribed (per DCI Corporate or local protocol or per physician on an individualized basis) must remain the same for at least 90 days prior to enrollment with respect to the ceiling for the total EPO dose administered per week, if a ceiling is used, and the level of hemoglobin (Hgb) at which EPO is discontinued (Hgb cutoff), if a Hgb cutoff is used.
4. The method by which IV Iron is prescribed (per DCI Corporate or local protocol or per physician on an individualized basis) must remain the same for at least 90 days prior to enrollment with respect to the serum ferritin and transferrin saturation (TSAT) targeted, if specific ferritin and TSAT targets are used

Exclusion Criteria:

1. Patients with a serum calcium ≥10.5 mg/dL on at least one occasion in the past 30 days.
2. Patients with a serum phosphorus >8.0 mg/dL on at least one occasion in the past 30 days.
3. Active infection defined by the use of IV antibiotic use within the past 30 days.
4. Current use of immunosuppressant medications other than low dose corticosteroids (prednisone <10 mg per day or equivalent)
5. History of a hematological malignancy (e.g. multiple myeloma, leukemia).
6. Sickle cell disease (sickle cell trait is not an exclusion).
7. Myelodysplasia requiring 1 or more blood transfusions in the past 3 months.
8. Transfusion for any reason within the past 30 days.
9. Medical conditions that cause a reduction in the absorption of oral vitamin D including Crohn's disease, celiac sprue, cystic fibrosis and surgical removal of part or all of the stomach or intestine.
10. Medications that cause a reduction in the absorption of oral vitamin D including cholestyramine (Questran, others), colestipol (Colestid, others) and orlistat (Xenical, Alli).
11. Known allergy/adverse reaction to ergocalciferol.
12. Treated with ergocalciferol and/or cholecalciferol (except if part of a multi-vitamin) within the last 3 months.
13. Average Kt/V < 1.3 on past three monthly labs. There must be at least 2 monthly Kt/V values in the past three months.
14. Skipped more than 3 dialysis treatments (excluding planned missed treatments) within the past 3 months for reasons other than hospitalization.
15. Life expectancy less than 6 months.
16. Kidney transplantation planned in the next 6 months.
17. Switch to peritoneal dialysis planned in the next 6 months.
18. Pregnant or planning to become pregnant within the next 6 months. A pre-menopausal woman must agree to use contraception for the duration of the study. If a woman has not had menses in over 12 months, consider this patient to be menopausal.
19. Unable or unwilling to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Actual)
Dates: Start 2011-06; Primary Completion 2014-04 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana Miskulin, MD, Principal Investigator — DCI
Locations (12):
- United States (12):
  - DCI - Redding, Redding, California
  - DCI - Albany, Albany, Georgia
  - DCI - Shreveport, Shreveport, Louisiana
  - DCI - Boston, Boston, Massachusetts
  - DCI- Columbia, Columbia, Missouri
  - DCI - Kansas City, Kansas City, Missouri
  - DCI- Omaha, Omaha, Nebraska
  - DCI - New Brunswick, New Brunswick, New Jersey
  - DCI - North Brunswick, North Brunswick, New Jersey
  - DCI - Philadelphia, Philadelphia, Pennsylvania
  - DCI - Knoxville, Knoxville, Tennessee
  - DCI - Maryville, Maryville, Tennessee

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 470 subjects were enrolled in the study; however 151 subjects did not make it to randomization due to EPO criteria not met n=45, did not meet other inclusion criteria n=57, no was reason provided n=49. Of the 319 subjects randomized, 43 had a baseline 25(OH)D >30. This analysis only pertains to the 276 subjects with a baseline 25(OH)D ≤30.
Period: Overall Study
Arm/Group | Ergocalciferol Supplementation | Placebo
Started | 137 | 139
Completed | 122 | 130
Not Completed | 15 | 9
Not completed — Death | 4 | 4
Not completed — Physician Decision | 3 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Transplant | 1 | 0
Not completed — GI symptoms | 1 | 0
Not completed — Withdrawal by Subject | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ergocalciferol Supplementation | Placebo | Total
Number analyzed (Participants) | 137 | 139 | 276
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (13.3) | 60.8 (13.9) | 61.1 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 58 | 125
  Male | 70 | 81 | 151
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 7 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 76 | 90 | 166
  White | 51 | 41 | 92
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 137 | 139 | 276
25Vit D (ng/mL) [Mean (Standard Deviation); unit: ng/mL] | 16.0 (5.9) | 16.9 (6.4) | 16.4 (6.2)
Epogen Dose, units/week [Median (Inter-Quartile Range); unit: units/week] | 5800 [2600 to 12200] | 5400 [2400 to 11500] | 5550 [2500 to 11900]

OUTCOME MEASURES:

1. Primary Outcome: EPO Dose
Description: The primary outcome is the change in the median EPO dose from baseline to 6 months after ergocalciferol supplementation.
Time Frame: Baseline, 6 months
Measure: Median (Inter-Quartile Range); unit: units/week
Arm/Group | Ergocalciferol Supplementation | Placebo
Number analyzed (Participants) | 122 | 130
units/week
  EPO dose - Baseline | 5800 [2600 to 12200] | 5400 [2400 to 11500]
  EPO dose - 6 months | 7000 [2500 to 16000] | 6050 [2000 to 11800]
Statistical Analysis 1: Comparison: Ergocalciferol Supplementation vs Placebo; Test type: Superiority or Other; p = 0.78, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Ergocalciferol Supplementation | Placebo
Serious Adverse Events (participants affected / at risk) | 4/137 | 4/139
Other Adverse Events (participants affected / at risk) | 9/137 | 8/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ergocalciferol Supplementation (N=137) | Placebo (N=139)
Death (Cardiac disorders) | 4 (4) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ergocalciferol Supplementation (N=137) | Placebo (N=139)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI agrees that the first publication and presentation shall be made by sponsor. If publication is not made within 24 months PI may publish their site data provided that sponsor receives 30 days to review.